CLINICAL TRIAL: NCT06984068
Title: Effect of Vitamin D Supplementation on the Rehabilitation of Patients After Rotator Cuff Tear Repair: a Double-blind Randomized Controlled Trial
Brief Title: Effect of Vitamin D Supplementation on the Rehabilitation of Patients After Rotator Cuff Tear Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Tim-Yun Michael ONG, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025.058
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Rotator Cuff Tear
Keywords: rotator cuff tear; rotator cuff tear repair; vitamin D
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive vitamin D supplement for 6 months
  Interventions: Drug: Vitamin D
- Control group (Placebo Comparator): The control group will receive placebo for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D — 4000IU/day vitamin D supplement will be used for 6 months
  Arms: Intervention group
Drug: Placebo — Placebo will be used for 6 months
  Arms: Control group

SUMMARY:
Rotator cuff tears are a significant health concern that severely affect shoulder joint mobility in patients. Common clinical manifestations of RCTs include shoulder pain, limited range of motion, joint instability, muscle weakness, and functional disability. In patients with rotator cuff tears, the prevalence of vitamin D deficiency ranges from 8.3% to 71%. Given its critical role in muscle strength and function, vitamin D is emerging as an important factor in the management of musculoskeletal disorders, including rotator cuff injuries. Despite the promising evidence regarding vitamin D's role in muscle strength and tendon healing, the specific impact of vitamin D supplementation on postoperative rehabilitation remains unclear. Given that vitamin D deficiency is easily diagnosed and treated, it is considered a modifiable risk factor that could be utilized in orthopedic care to improve patient outcomes. Vitamin D supplementation is a cost-effective and potentially efficient intervention that may enhance muscle strength, reduce postoperative pain, and improve joint function in patients recovering from rotator cuff repair. The objective of this study is to investigate the effects of vitamin D supplementation on postoperative outcomes in patients undergoing arthroscopic rotator cuff repair. The study will be conducted as a randomized controlled trial, with participants receiving either a daily dose of 4000 IU of vitamin D or a placebo. The primary outcomes to be evaluated include muscle strength, postoperative pain, and joint function. Blood samples will be collected at baseline, and after 3 months, 6 months, and 12 months of supplementation to monitor the effects of vitamin D on serum levels and its correlation with clinical outcomes.

DETAILED DESCRIPTION:
Rotator cuff tears is one of the diseases that severely affect the movement of the shoulder joint in patients. The clinical manifestations of rotator cuff tears typically include shoulder pain, restricted range of motion, joint instability, muscle weakness, and functional disability. Epidemiological data reveal a progressive increase in the prevalence of rotator cuff injuries among middle-aged and older adults. The prevalence is estimated to be approximately 15-20% in individuals aged 60 years, 26-30% in those aged 70 years, and up to 50% in individuals aged 80 years.

Risk factors for rotator cuff tears are multifactorial, including age, smoking, hypercholesterolemia, history of trauma or repetitive overhead activity, dominant arm injury, and family history of shoulder problems. The wide variation in the causes of rotator cuff tears, coupled with the prevalence of asymptomatic tears, has contributed to a lack of standardization in treatment approaches. While physical therapy and regenerative medicine treatments, such as platelet-rich plasma (PRP) and stem cell therapy, have been explored as potential alternatives, evidence suggests that the intrinsic healing capacity of the rotator cuff is limited. Arthroscopic rotator cuff repair is considered the treatment of choice for acute tears across all age groups, as well as for patients under the age of 65 with chronic, large (>1 cm), reparable tears and no irreversible muscle changes. Despite advancements in surgical techniques, the rehabilitation process remains challenging due to the biomechanical complexity of the shoulder and the multifactorial nature of recovery. Many patients experience suboptimal outcomes, including muscle weakness, persistent pain, functional limitations, and re-tearing of the rotator cuff.

Vitamin D insufficiency or deficiency is widely recognized as being closely associated with the development of various conditions, including osteoporosis, fractures, and muscle weakness. It is estimated that up to 32% of the U.S. population and as many as one billion people worldwide are affected by Vitamin D deficiency or insufficiency (defined as a 25(OH)D3 level >20 ng/mL but <30 ng/mL). The prevalence of Vitamin D deficiency is notably high among orthopedic patient populations. A retrospective study revealed that 43% of patients undergoing preoperative evaluation exhibited Vitamin D insufficiency, with 40% classified as deficient. Vitamin D deficiency prevalence ranges from 8.3% to 71% in patients with rotator cuff tears. Vitamin D's impact on muscle strength and function has made it a subject of increasing interest in the management of musculoskeletal disorders, including rotator cuff injuries.

Current research on rotator cuff injuries has indicated a potential role for vitamin D in enhancing tendon healing. By inhibiting matrix metalloproteinases (MMPs), which hinder rotator cuff repair, vitamin D facilitates the accumulation of fibrocartilage and collagen, thereby improving tendon healing. Animal experiments have shown that vitamin D supplementation can enhance muscle fiber size, improve muscle function, reduce the expression of pro-fibrotic genes, and increase the expression of anti-fibrotic genes. This, in turn, helps mitigate muscle fatty infiltration and improve skeletal muscle quality regulation signaling pathways. One study reported through regression analysis that serum vitamin D levels were significantly negatively correlated with rotator cuff fatty degeneration. Furthermore, another study conducted muscle biopsies on patients undergoing rotator cuff repair and compared those deficient in vitamin D with patients who had sufficient levels. They found significantly increased expression of pro-inflammatory genes IL1β and IL6 in the deltoid and supraspinatus muscles of vitamin D-deficient individuals. This heightened postoperative inflammatory response may delay muscle repair and functional recovery, leading to suboptimal rehabilitation outcomes. Low vitamin D concentrations may serve as an independent variable contributing to fatty infiltration and degeneration of the supraspinatus and infraspinatus muscles. Another study demonstrated a significant association between low preoperative vitamin D levels and increased complications following rotator cuff repair. In patients undergoing arthroscopic rotator cuff repair, lower vitamin D levels were correlated with more severe muscle weakness at one year postoperatively. Additionally, preoperative vitamin D deficiency has been linked to higher re-tear rates and increased early postoperative pain.

Despite the promising evidence, the specific role of vitamin D in postoperative rehabilitation remains unclear. Given the ease of diagnosis and treatment of vitamin D deficiency, it is considered a highly modifiable risk factor in orthopedic care. Vitamin D supplementation holds promise as a cost-effective and efficient intervention that may improve postoperative outcomes, including enhanced muscle strength and joint function, in patients undergoing rotator cuff repair. Therefore, this study aims to investigate the effects of vitamin D supplementation on postoperative outcomes in patients undergoing arthroscopic rotator cuff repair. Using a randomized controlled trial (RCT) design, this study will evaluate the impact of vitamin D supplementation on muscle strength, postoperative pain, and joint function in patients with rotator cuff tears.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged between 40 and 70 years.
2. Clinically and radiologically (magnetic resonance imaging) diagnosed full-thickness supraspinatus tendon tears that were confirmed by arthroscopic surgery and could be surgically repaired.
3. Degree of supraspinatus tendon tear according to the DeOrio and Cofield grading system as moderate tear (1-3 cm) and mild tear (<1 cm).
4. Serum vitamin D level <30 ng/mL >20 ng/mL before rotator cuff tears surgery
5. Signed informed consent and underwent 12-month follow-up.

Exclusion Criteria:

1. Presence of other shoulder pathologies such as subscapularis tear, adhesive capsulitis, long head of biceps tendonitis, calcific tendonitis, or shoulder tumor.
2. Large or unrepairable rotator cuff tear (>3 cm).
3. Previous history of shoulder surgery or recurrent rotator cuff tears.
4. Combined injury to the shoulder labrum, articular cartilage or biceps tendon.
5. Contraindications to vitamin D supplementation (e.g., allergies).
6. Serious comorbidities such as cardiovascular disease.
7. Severe osteoporosis or rheumatoid arthritis.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
External and internal rotation isometric strength of the shoulder | Baseline, 3 months, 6 months and 12 months post-intervention
  Isometric shoulder strength will be tested using an isokinetic dynamometer (Biodex System 2, Shirley, New York). Following the protocol described by Hughes and colleagues, strength testing will be performed at the following joint positions: coronal-plane abduction (ABD) at 30° of abduction, internal rotation (IR) at 15° of frontal-plane elevation and 0° of humeral rotation, and external rotation (ER) at 15° of frontal-plane elevation and 0° of humeral rotation. To isolate shoulder strength and minimize the likelihood of compensation with other muscle groups, patients will be secured to the Biodex system with 2 hook-and-loop straps diagonally across their torso. Three trials will be performed at each position, with at least 2 minutes of rest between each trial. The average of the 3 trials will be calculated and recorded as the patient's maximum isometric strength. Both shoulders will be tested, and the testing order will be randomized. To account for any inherent differences in strengt

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline, 3 months, 6 months and 12 months post-intervention
  The VAS is used for determination of the pain intensity. The VAS scale is represented as a 10 cm-long line. The left side of the line (0) corresponds to "no pain" and the right side (10) represents "the worst pain ever"
the American Shoulder and Elbow Surgeons (ASES) score | Baseline, 3 months, 6 months and 12 months post-intervention
  The ASES questionnaire is used for evaluation. The ASES score consists of two subscales: activities of daily living (ADL) and pain. It is a patient-reported outcome measure, ranging from 0 (severe pain and complete loss of function) to 50 (no pain and good function) for each subscale. The total score is obtained by summing the two subscale scores, with a maximum possible score of 100 points
the University of California, Los Angeles (UCLA) score | Baseline, 3 months, 6 months and 12 months post-intervention
  The UCLA Shoulder Score is a widely used scale for evaluating shoulder function following rotator cuff repair. It primarily assesses shoulder pain, function, range of motion, and patient satisfaction with the outcomes of shoulder treatment
the Constant-Murley score | Baseline, 3 months, 6 months and 12 months post-intervention
  The Constant-Murley Score, introduced by Constant and Murley, is another commonly used questionnaire for shoulder assessment. It evaluates various aspects of shoulder function, including range of motion, strength, and overall functionality. The range of motion assessment is comprehensive, covering forward flexion, external rotation, abduction, and internal rotation. The total score ranges from 0 to 100, with higher scores indicating better shoulder function
Range of motion (ROM) | Baseline, 3 months, 6 months and 12 months post-intervention
  ROM is measured using a goniometer and includes forward flexion (anterior elevation in the sagittal plane), abduction (posterolateral elevation in the coronal plane), external rotation (forearm abduction of 90° with outward rotation), and internal rotation (arm abduction of 90° with extension behind the back or inward rotation). The test will be repeated twice and the mean values will be analyzed
Magnetic resonance imaging (MRI) | Baseline, 12 months post-intervention
  Magnetic resonance imaging (MRI) was performed on all patients, including coronal, sagittal, and axial T2-weighted echo scans. Tendon integrity was classified according to Sugaya et al. into five types. Type I describes an intact tendon with normal thickness and uniform signal. Type II corresponds to an intact tendon with normal thickness but increased internal signal. Type III describes a repaired tendon with a thickness reduced by up to 50% compared to a healthy tendon, with increased internal signal. Type IV represents a partial rupture, and Type V represents a complete rupture or lack of tendon integration. Atrophy of the supraspinatus muscle was assessed at the "Y-shaped" view on the T1-weighted sagittal cut that included both the scapular spine and the corocoid using a tangent sign. The tangent sign is positive for atrophy if the superior border of the supraspinatus muscle is below a line drawn from the superior aspects of the scapular spine and corocoid.
Serum vitamin D assays | Baseline, 12 months post-intervention
  Blood samples will be taken under non-fasting conditions. Blood samples will be collected four times: Blood samples will be collected four times: before Vitamin D supplementation, at 3 months of supplementation, at 6 months of supplementation, and 6 months after the intervention. Each time, 5 ml of blood will be collected. Serum / plasma obtained will be immediately stored at -80°C until analysis. Serum 25 (OH) Vit-D assay: Serum 25 (OH) Vit-D levels will be measured by commercial 25 (OH) Vitamin D ELISA kit (Abcam ab213966) according to the manufacturer's instruction, providing the quantitative determination of 25 (OH) Vitamin D3 and 25 (OH) Vitamin D2. Sensitivity: 1.98 ng/ml (Range: 0.5 ng/ml - 1010 ng/ml).

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 6 months after publication
Access Criteria: Journal reviewer